CLINICAL TRIAL: NCT00944320
Title: Pharmacogenetics of Antifolate Disease Modifying Anti-Rheumatic Drugs in Rheumatoid Arthritis in Taiwan
Status: Completed | Type: Observational
Sponsor: National Chung Hsing University (Other)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: En-Pei Isabel Chiang, Department of Food Science and Biotechnology of National Chung Hsing University
Other Study IDs: C05133
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Polymorphisms occur in several genes encoding key enzymes in the folate pathway may affect drug metabolism in patients with rheumatoid arthritis. Whether these genetic variations contribute to differential responses to antifolate drug in patients with rheumatoid arthritis (RA) remains to be investigated in the Taiwanese population.

Objective. The goal of the present study is to investigate the interactions between genetic variations in folate genes and the efficacy/side effects of anti-folate disease-modifying antirheumatic drug in Taiwan.

DESIGN. A cross-sectional study involving 100 patients with RA were enrolled from TCVGH. Genotypes in methylenetetrahydrofolate reductase (MTHFR677C>T), tandem repeat polymorphism in thymidylate synthase enhancer region (TSER) and folylpoly-gamma-glutamate synthetase (FPGS1901T>C) were determined by RFLP or pyrosequencing.

ELIGIBILITY:
Inclusion Criteria:

* Male/female age >18
* Clinical diagnosis of Rheumatoid Arthritis

Exclusion Criteria:

* Must not be pregnant/breastfeeding
* Other conditions may lead to exclusion from the trial (e.g. Diabetes mellitis, malignant melanoma, cardiac conduction disorders, hepatic/renal insufficiency.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cross-sectional study involving 100 patients with RA were enrolled from TCVGH.
Sampling Method: Probability Sample
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)